CLINICAL TRIAL: NCT04886388
Title: Open-Label, Randomized, Controlled, Parallel-Group Trial of a Digital Therapeutic for the Treatment of Type 2 Diabetes
Brief Title: Pivotal Trial of a Digital Therapeutic for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Better Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM2-06
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized, Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BT-001 + Standard of Care (Experimental): BT-001 is a software program used with physician guidance, being investigated to improve glycemic control. Patients randomized to this arm of the study will interact with the BT-001 software program in addition to receiving Standard of Care for type 2 diabetes
  Interventions: Device: BT-001; Other: Physician-guided Standard of Care for type 2 diabetes
- Standard of Care (Active Comparator): Patients randomized to the Standard of Care arm will receive Standard of Care treatment for type 2 diabetes under the guidance of a physician
  Interventions: Other: Physician-guided Standard of Care for type 2 diabetes

INTERVENTIONS:
Device: BT-001 — BT-001 is a software program intended to help patients with type 2 diabetes, under the guidance of their physician, improve glycemic control.
  Arms: BT-001 + Standard of Care
Other: Physician-guided Standard of Care for type 2 diabetes — Current ADA Standard of Care Guidelines for type 2 diabetes

SUMMARY:
BT-001 is a software program intended to help patients with type 2 diabetes, under the guidance of their physician, improve glycemic control (i.e., levels of blood sugar). The BT-001 software delivers a type of behavioral therapy to patients via a mobile application that targets behaviors related to achieving glycemic control. The effectiveness of BT-001 will be measured by its ability to help patients reduce Hemoglobin A1c, or HbA1c (a marker in the blood that measures blood sugar) compared to standard medical care in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The study will utilize an open-label, randomized, parallel-group design to confirm and characterize the safety and efficacy of BT-001 used in addition to standard of care (SOC) when compared to SOC alone in patients with type 2 diabetes. The screening period will consist of a run-in during which time HbA1c will be assessed for confirmation of eligibility.

Once confirmed to be eligible, patients will then be randomized 1:1 to the following groups:

Investigational: One half of the participants will be treated with BT-001 plus SOC for 180 days;

Control: One half of the participants will be treated with SOC alone for 180 days.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years old, inclusive at the time of signing the informed consent;
2. Diagnosis of type 2 diabetes, according to the criteria of the American Diabetes Association (ADA), and confirmed at the initial eligibility screening;
3. Body Mass Index ≥25 kg/m2;
4. Possesses a smartphone (iPhone or Android only) capable of running the smartphone applications (Apps) used in the study;
5. Has had no change in the last 4 months prior to randomization (3 months prior to initial screening plus 30-day run-in screening period) in antihyperglycemic medications;
6. Has a current HbA1c level >7%, as determined by both screening assessments;
7. Willing to use an FDA approved glucometer for self-monitoring blood glucose throughout the study;
8. Is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria

1. Are unable to understand, consent to, or comply with the study protocol for any reason;
2. Currently taking prandial (mealtime) insulin;
3. Have self-reported measures, collected during screening interview, that reveal:

   1. An active eating disorder
   2. The taking of or planning to take (within the next 6 months):

   i. Oral steroids (planned, or within the past 3 months) ii. Chemotherapy (planned, or within the past 6 months) iii. Weight loss medications or iv. Atypical antipsychotic medications

   c. A change in antidepressant or anti-anxiety medication within the past 3 months;

   d. A history of bariatric surgery or planned bariatric surgery during the study;

   e. The current use of marijuana, cocaine, opioid painkillers, or other addictive substances;

   f. The current use of tobacco products or use of tobacco products within the past 6 months;

   g. The consumption of alcohol above defined thresholds:

   i. For women: more than 3 drinks in a single day, or more than 7 drinks per week and ii. For men: more than 4 drinks in a single day, or more than 14 drinks per week

   h. An unstable or life-threatening medical illness;

   i. Non-resolved, presumed or confirmed COVID-19 diagnosis prior to randomization or during primary study period;

   j. For women only: pregnant (or lactating) or having the intention of becoming pregnant during the time frame of the study.
4. Has a current HbA1c level ≥11%, at the screening assessment;
5. Concurrent enrollment in any other clinical trial;
6. Is considered unreliable by the investigator, or having any condition which, in the opinion of the investigator, would not allow safe participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
The difference in the mean change from baseline in HbA1c at Day 90 between Intervention and Standard of Care groups | Baseline and Day 90
  Hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin.

SECONDARY OUTCOMES:
The difference in the mean change from baseline in HbA1c at Day 180 between Intervention and Standard of Care groups | Baseline and Day 180
  Hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berman, MD, Study Director — Better Therapeutics
Locations (6):
- United States (6):
  - Study Site, San Francisco, California
  - Study Site, Miami, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Chicago, Illinois
  - Study Site, New York, New York
  - Study Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No